CLINICAL TRIAL: NCT00261105
Title: An Open, Multicenter, Non-comparative, Phase IV Trial of Efficacy and Safety of Ketek(Telithromycin) 800mg
Brief Title: Telithromycin in Respiratory Tract Infections
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMR3647A_4026
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections | interventions — telithromycin

INTERVENTIONS:
Drug: telithromycin

SUMMARY:
Primary Objectives:

* The primary objective of the study is to evaluate clinical efficacy i.e. to show that with respect to clinical cure rate, Ketek® (telithromycin) in the treatment of community acquired respiratory tract infections: community acquired pneumonia (CAP), acute bacterial exacerbation of chronic bronchitis (AECB) and acute sinusitis (AS), in outpatients.

Secondary Objectives:

The secondary objectives are to:

* Further assess the efficacy of Ketek® (telithromycin) by considering the rate at which additional antibacterials were prescribed to treat the primary infection; the rate of hospitalisation due to a complication of the primary infection and assessment of bacteriological data, chest X-ray and sinus X-ray if available.
* Evaluate safety of Ketek® (telithromycin) through Adverse Event (AE) and Serious Adverse Event (SAE) reporting

ELIGIBILITY:
Inclusion Criteria:

General Conditions

* Outpatients
* Fulfillment of clinical diagnostic criteria for one of the following indications:

  * Mild to moderate Community Acquired Pneumonia (CAP)
  * Acute bacterial Exacerbation of Chronic Bronchitis (AECB)
  * Acute Sinusitis (AS)

For CAP

The Criteria to be fulfilled are:

* New onset of at least two of the following:

  * Cough
  * Production of purulent sputum
  * Auscultatory findings compatible with pneumonia, e.g. rales, evidence of pulmonary consolidation
  * Dyspnea or tachypnea
  * Fever
  * Elevated total white blood cell count > 10 000/mm3 or >15% bands regardless of total count
* Chest X-ray findings supporting a clinical diagnosis of bacterial pneumonia (e.g. new infiltrate)

For AECB

The Criteria to be fulfilled are:

* Chronic bronchitis defined as cough and excessive sputum production for more than 2 consecutive years and on most days in a 3-month consecutive period.
* Exacerbation defined by:

  * Increase in sputum purulence, or
  * Increase in sputum volume, or
  * Increase in dyspnea

For AS

The criteria to be fulfilled are:

At least two of the major or one major and two minor factors listed below, for more than one week and less than 4 weeks:

* Major factors:

  * Facial pressure and/or pain
  * Facial congestion or fullness
  * Nasal obstruction
  * Nasal purulence or postnasal discharge
  * Hyposmia or anosmia
  * Fever
* Minor factors:

  * Headache
  * Halitosis
  * Fatigue
  * Dental pain
  * Cough
  * Ear pain, pressure or fullness

Exclusion Criteria:

General Conditions

Subjects presenting with any of the following will not be included in the study:

* Treatment required during the study with ergot alkaloid derivatives, pimozide, astemizole, terfenadine, cisapride, simvastatin, atorvastatin and lovastatin, and the oral use of the benzodiazepines midazolam, triazolam and alprazolam.
* History of congenital or family history of long QT syndrome (if not excluded by ECG) or known acquired QT interval prolongation.
* Known hypersensitivity to telithromycin or to macrolide antibiotics.
* Hospital acquired infections (hospitalization for more than 72 hours within 7 days of study entry).
* Pregnant or breast-feeding women. For the women of childbearing potential it is left to the investigators discretion to establish a lack of pregnancy, e.g. with contraceptive use, menstrual pattern, urinary pregnancy test.
* Subjects with severely impaired renal function (creatinine clearance <30 ml/min).
* Subjects that had received anti-bacterials for more than 24 hours within 7 days prior to enrollment in the study, unless the treatment has failed.
* Subjects receiving medications, including other anti-microbials or anti-cancer drugs, that could interfere with the evaluation.
* Microbiologically documented infection with a pathogen known prior to inclusion to be resistant to the study medications.
* Infection, other than the primary infection for which the subject is being included in the study that requires use of other systemic anti-bacterial drug.
* Splenectomised subjects.
* Use of Ketek® (telithromycin) or participation in a study using Ketek® (telithromycin) in the previous 30 calendar days.
* Subjects that have received any investigational drug within 4 weeks of enrollment in the study.
* No subject will be allowed to enroll in this study more than once.

For CAP

Additional exclusion criteria are:

* Severe pneumonia defined by any one of the following:

  * Judged as needing Intensive Care Unit admission.
  * Need of parenteral antibiotic treatment (if the attending physician wants to prescribe a parenteral treatment for adherence reasons or local prescription habits this is accepted, provided that the patient does not have a severe pneumonia).
  * Acute respiratory failure or requirement for mechanical ventilation.
  * Altered mental status resulting from the infective process.
  * Resting respiratory rate > 30 breaths/min.
  * Chest X-ray showing increase in opacity by > 50% within 48 hours of current evaluation.
* Total white blood cell count < 4 000/mm3.
* Aspiration pneumonia.
* Pneumonia suspected to be non-bacterial (due to fungus or viral).
* Subjects suffering from severe bronchiectasis (production of more than 125 mL of sputum/day), cystic fibrosis, active tuberculosis, pulmonary infarction or embolism, bronchial obstruction, lung cancer or lung metastasis, lung abscess, extra-pulmonary extension (like meningitis, septic arthritis, endocarditis).

For AECB

Additional exclusion criteria are:

* Need of parenteral antibiotic treatment (if the attending physician wants to prescribe a parenteral treatment for adherence reasons or local prescription habits this is accepted, provided that the patient does not have a severe infection).
* Acute respiratory failure (respiratory distress, hypercarbia, worsening hypoxemia) or requirement for mechanical ventilation.
* Severe bronchiectasis, cystic fibrosis, active tuberculosis, pulmonary infarction or embolism, bronchial obstruction, lung cancer or lung metastasis, lung abscess.

For AS

Additional exclusion criteria are:

* Need of immediate surgery for the treatment of AS.
* Chronic sinusitis (symptoms lasting more than 4 weeks).
* Recurrent sinusitis (4 or more episodes of sinusitis requiring antibiotic therapy in the previous 12 months).
* Nosocomial acquired sinusitis.
* Cystic fibrosis, immotile cilia syndrome.
* Obstructive lesions in nasopharynx (e.g. polyps, tumor).
* Use of nasal, nasogastric or nasotracheal catheters.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-02; Primary Completion 2005-10 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome (Global Assessment by the participating physicians) | During the Study Conduct

SECONDARY OUTCOMES:
Rate at which additional antibacterials were prescribed to treat the primary infection | During the study conduct
Rate of hospitalisation due to a complication of the primary infection | During the study conduct
Assessment of chest X-ray and sinus X-ray if available. | During the study conduct
Adverse Event (AE) and Serious Adverse Event (SAE) reported | from the inform consent signed up to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Won-Sik Lee, MD, Study Director — Sanofi